CLINICAL TRIAL: NCT06286527
Title: Quality of Sexual Life of PrEP Users
Acronym: PREP-QUAL-VS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: EssaiClinique_PREP-QUAL-VS
Record Dates: First submitted 2024-01-18; First posted 2024-02-29 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: HIV Pre-exposure Prophylaxis Use; Adult
Keywords: PrEP (HIV pre-exposure prophylaxis); quality of life; sexual life

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult PrEP users
  Interventions: Other: anonymous self-administered online questionnaire

INTERVENTIONS:
Other: anonymous self-administered online questionnaire — proposition to participate through billboards with a QR code leading to the questionnaire.

SUMMARY:
The study will recruit participants on the occasion of their visit in a sexual health center or another HIV pre-exposure prophylaxis (PrEP) facility in France.

PrEP users will be proposed to fill a self-administered, online, anonymous questionnaire regarding how they perceive different fields of their sexual life, and how they perceive that PrEP has an impact on the quality of sexual life.

DETAILED DESCRIPTION:
PrEP aims to protect against HIV; more broadly, PrEP is a holistic process, addressing vaccination (hepatitis A, hepatitis B, human papillomavirus, MPox), sexually transmitted infection diagnosis, mental health, issues related to psychoactive substance use, etc.

This process is likely to impact not only "classical" health areas, but also fields concerning more widely the quality of life.

In particular, the investigators emit the hypothesis that PrEP is associated with an increase of the quality of sexual life.

the investigators have therefore designed a study based on a self-administered anonymous questionnaire to explore how PrEP user evaluate their quality of sexual life and how they perceive the impact of PrEP on this topic.

Adult PrEP users will be recruited through billboard in sexual health center or another PrEP facility in France. A QR (quick response) code will be displayed, giving access to the questionnaire.

Participation to the study is limited to fill once the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* current PrEP use
* adult

Exclusion Criteria:

* unwilling to participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: current PrEP users in sexual health centers or other PrEP facilities
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-09-06 (Estimated); Study Completion 2024-09-06 (Estimated)

PRIMARY OUTCOMES:
quality of sexual life as assessed by a set of questions | inclusion
  The study relies on a self-administered, online, anonymous questionnaire of 40 questions. Some of these questions will allow assessing the perceived quality of sexual life, by exploring if participants are satisfied with the number of their partners, the sexual intercourses they have, the orgasms they reach, the lack of anxiety during mating and sexual intercourse, the bond they create with their partner(s), the feeling of fulfilment they have regarding their sexual intercourses. THE ANSWERS TO THE DATA WILL NOT BE USED TO CREATE A NUMERICAL SCALE.
perceived influence of PrEP use on the quality of sexual life | inclusion
  Some questions of the already mentioned self-administered, online, anonymous questionnaire will allow assessing the perceived link between PrEP and quality of sexual life. More precisely, Participants will be asked the extent to which they see a link between PrEP use and the perceived quality of their sexual life in different axes (physical, emotional).

CONTACTS AND LOCATIONS:
Locations (1):
- Olivier EPAULARD, Grenoble, Is, France

IPD SHARING:
Plan to Share IPD: No